CLINICAL TRIAL: NCT03620526
Title: Inhaled Iloprost and Exercise Hemodynamics and Ventricular Performance in Heart Failure With Preserved Ejection Fraction - the ILO-HOPE Clinical Trial
Brief Title: Inhaled Iloprost and Exercise Hemodynamics and Ventricular Performance in Heart Failure With Preserved Ejection Fraction
Acronym: ILO-HOPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201704075MIND
Record Dates: First submitted 2018-06-21; First posted 2018-08-08 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Iloprost; Heart failure with preserved ejection fraction; hemodynamic; Pulmonary wedge pressure
MeSH Terms: interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iloprost (Experimental): patients received inhaled iloprost 10 mcg/mL x 1 dose after baseline and exercise test and then received measurements for hemodynamic data again for both baseline and after exercise test.
  Interventions: Drug: Iloprost
- Placebo (Placebo Comparator): patients received inhaled normal saline with the same amount x 1 dose after baseline and exercise test and then received measurements for hemodynamic data again for both baseline and after exercise test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloprost — Investigators performed cardiac catheterization as previously described. Hemodynamic values were recorded for the ﬁrst exercise phase (before any drug administration) and after return to steady state baseline hemodynamic values, and the second exercise phase (after drug administration). Subjects were randomized 1:1 to inhalation of placebo (normal saline solution) or iloprost (50 mg/kg/min) (Bayer Pharmaceuticals, Scottsdale, Ari-zona) for 5 min. The iloprost/placebo inhalation were identical in appearance and prepared by the research pharmacy, ensuring double-blinding of inhalation content. After finishing inhalation process for 10 min, hemodynamic measurements were repeated at rest, followed by repeat supine exercise at a 20-W workload for 6 min, identical to the study's ﬁrst phase.
  Arms: Iloprost
Drug: Placebo — Investigators performed cardiac catheterization as previously described. Hemodynamic values were recorded for the ﬁrst exercise phase (before any drug administration) and after return to steady state baseline hemodynamic values, and the second exercise phase (after drug administration). Subjects were randomized 1:1 to inhalation of placebo (normal saline solution) or iloprost (50 mg/kg/min) (Bayer Pharmaceuticals, Scottsdale, Ari-zona) for 5 min. The iloprost/placebo inhalation were identical in appearance and prepared by the research pharmacy, ensuring double-blinding of inhalation content. After finishing inhalation process for 10 min, hemodynamic measurements were repeated at rest, followed by repeat supine exercise at a 20-W workload for 6 min, identical to the study's ﬁrst phase.
  Arms: Placebo

SUMMARY:
BACKGROUND There is no effective medical treatment for heart failure with preserved ejection fraction (HFpEF). Increases in pulmonary capillary wedge pressure (PCWP) develop in patients with HFpEF. Prostacyclin analogo can possible reduced PA pressure along with PWCP pressure, as with exercise.

OBJECTIVES This study try to determine whether inhlalation of iloprost improves exercise hemodynamics and cardiac reserve in HFpEF.

METHODS In a double-blind, randomized, placebo-controlled, parallel-group trial, subjects with HFpEF underwent invasive cardiac catheterization with simultaneous expired gas analysis at rest and during exercise, before and 15 min after treatment with either inhaled iloprost or matching placebo.

DETAILED DESCRIPTION:
Study participants and study design The ILO-HOPE trial is a prospective, randomized, double-blind, single center trial conducted at the National Taiwan University Hospital (NTUH). This study was performed in accordance with the Declaration of Helsinki and was approved by the institutional review board of the National Taiwan University Hospital, and all subjects provided their written informed consent prior to participation in the study. Patients referred to National Taiwan University Hospital cardiac catheterization laboratory for invasive hemodyanamic exercise stress testing were enrolled. HFpEF was defined according to 2016 European society of cardiology heart failure guidelines and our previous studies. In brief, HFpEF was determined by (1) presence of typical HF symptoms and signs (2) LV ejection fraction ≥ 50 (3) elevated levels of NT-proBNP (at least >125 pg/ml) (4) echocardiographic structural (a left atrial volume index > 34 mL/m2 or a left ventricular mass index ≥115 g/m2 for males and ≥95 g/m2 for females) or functional alterations (E/e'≥13 and a mean e' septal and lateral wall < 9 cm/s). The exclusion criteria were chronic renal failure (creatinine > 250 μmol/L), significant hepatic disease, secondary hypertension, pericardial disease, valvular heart disease (echocardiographic evidence of at least mild stenosis or at least moderate regurgitation), cancer, cor pulmonale, congenital heart disease, left-to-right shunt, myocardial infarction within 60 days, high-output heart failure, long-term treatment with phosphodiesterase 5 inhibitors, and chronic atrial fibrillation. The patients will be asked to hold nitrate for 3 days before the test if they receive any oral nitrate.

Trial protocol Investigators will perform cardiac catheterization with simultaneous expired gas analysis at rest and during supine exercise at a 20-W workload for 6 min, as previously described. Hemodynamic values will be recorded for the ﬁrst exercise phase (before any drug administration) and after return to steady state baseline hemodynamic values, and the second exercise phase (after drug administration). Subjects will be randomized 1:1 to inhalation of placebo (normal saline solution) or iloprost (50 mg/kg/min) (Bayer Pharmaceuticals, Scottsdale, Ari-zona) for 5 min. The iloprost/placebo inhalation will be identical in appearance and prepared by the research pharmacy, ensuring double-blinding of inhalation content. After finishing inhalation process for 10 min, hemodynamic measurements will be repeated at rest, followed by repeat supine exercise at a 20-W workload for 6 min, identical to the study's ﬁrst phase. Arterial and venous blood samples and hemodynamic and expired gas data will be acquired during each stage of the protocol. Right heart catheterization will be performed through a 7-F sheath via the internal jugular vein. Transducers were zeroed at mid-axilla. Right atrial pressure (RAP), pulmonary artery (PA) pressure, and PCWP will be measured at end-expiration using swan-Ganz catheter 2-F, high-ﬁdelity micromanometer-tipped cathe-ters (Millar Instruments, Houston, Texas) advanced through the lumen of a 7-F, ﬂuid-ﬁlled catheter (Arrow, Teleﬂex, Morrisville, North Carolina)(). Mean RAP and PCWP will be taken at mid A wave. Arterial blood pressure (BP) will be measured continuously through a 5-F radial arterial cannula. Oxygen consumption (VO2) will be measured from expired gas analysis (MedGraphics, St. Paul, Minnesota) taken as the average from the 60 s preceding arterial and mixed venous blood sampling. Ventilatory efﬁciency will be assessed by the increase in minute ventilation relative to carbon dioxide production (VE/VCO2). CO and stroke volume (SV) will be determined by the direct Fick method and heart rate as previous described. Investigators also will calculate pulmonary vascular resistance, PA compliance (SV/PA pulse pressure), and systemic vascular resistance (SVR) using standard formulas. LV systolic performance will be assessed by LV stroke work using standard formula as well.

Assessments of outcomes The primary endpoint of the trial is the PCWP during exercise. Secondary endpoints are changes of other hemodynamic data including alterations in resting PCWP, rest and exercise changes in RAP, PA pressure, PVR, PA compliance, systemic BP, heart rate, SV, stroke work.

Statistical analysis Statistical analyses will be done on an intention to treat basis. Results are reported as mean ± SD, median (interquartile range) or n (%).Within-group differences are assessed by the paired Student t test. Between-group differences in rest or exercise hemodynamic responses were compared by an unpaired Student t test., Wilcoxon rank sum test, or Fisher exact test. Linear regression will be performed to compare hemodynamic responses to exercise before and after study drug inhalation, with variables log-transformed as necessary for analysis. All tests were 2-sided, with p < 0.05 considered signiﬁcant. We used G-power (version 3.1.9.2, Heinrich-Heine-Universität Düsseldorf, Germany; http://www.gpower.hhu.de/) to calculate the sample size. A sample size of 34 total patients would be needed to provide 80% power (assuming a SD of 2.76 mmHg) to detect a 2 mmHg difference in the primary efficacy parameter, change in exercising PCWP, with a 5% type I error rate for a 2-sided test.

ELIGIBILITY:
Inclusion Criteria:

1. presence of typical HF symptoms and signs
2. LV ejection fraction ≥ 50
3. elevated levels of NT-proBNP (at least >125 pg/ml)
4. echocardiographic structural (a left atrial volume index > 34 mL/m2 or a left ventricular mass index ≥115 g/m2 for males and ≥95 g/m2 for females) or functional alterations (E/e'≥13 and a mean e' septal and lateral wall < 9 cm/s).

Exclusion Criteria:

1. chronic renal failure (creatinine > 250 μmol/L)
2. significant hepatic disease, significant coronary artery disease (CAD) (coronary artery stenosis >70% without intervention or positive stress test),
3. secondary hypertension,
4. pericardial disease
5. significant valvular heart disease (>mild stenosis, >moderate regurgitation),
6. active cancer,
7. cor pulmonale
8. congenital heart disease
9. high-output heart failure
10. subjects receiving long-term treatment with phosphodiesterase 5 in-hibitors
11. chronic atrial fibrillation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary wedge pressure changes after exercise measured by swan-ganz catheter (effect of inhalation of drug[efficacy]) | 15 minutes after inhalation of drugs
  Exercise pulmonary wedge pressure changes measured by swan-ganz catheter

SECONDARY OUTCOMES:
Resing pulmonary wedge pressure measured by swan-ganz catheter (effect of inhalation of drug[efficacy]) | 15 minutes after inhalation of drugs
  resting pulmonary wedge pressure changes measured by swan-ganz catheter
Resting cardiac output as assessed by direct Fick method and heart rate (effect of inhalation of drug[efficacy]) | 15 minutes after inhalation of drugs
  Investigators will measured cardiac output by direct Fick method and heart rate before exercise, after exercise, after inhalation of drugs(placebo/iloprost) and after second exercise. The outcomes will be the absolute value of cardiac output at rest before and after inhalation of the different drug.
Resting pulmonary vascular resistance as assessed by direct Fick method and heart rate (effect of inhalation of drug[efficacy]) | 15 minutes after inhalation of drugs
  Investigators will measured cardiac output and also pulmonary vascular resistance by direct Fick method and heart rate before exercise, after exercise, after inhalation of drugs(placebo/iloprost) and after second exercise. The outcomes will be the absolute value of pulmonary vascular resistance at rest before and after inhalation of the different drug.

CONTACTS AND LOCATIONS:
Overall Officials: CHO-KAI WU, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Borlaug BA, Koepp KE, Melenovsky V. Sodium Nitrite Improves Exercise Hemodynamics and Ventricular Performance in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2015 Oct 13;66(15):1672-82. doi: 10.1016/j.jacc.2015.07.067. PMID 26449137
- [Derived] Chen ZW, Huang CY, Cheng JF, Chen SY, Lin LY, Wu CK. Stress Echocardiography-Derived E/e' Predicts Abnormal Exercise Hemodynamics in Heart Failure With Preserved Ejection Fraction. Front Physiol. 2019 Dec 3;10:1470. doi: 10.3389/fphys.2019.01470. eCollection 2019. PMID 31849715
- [Derived] Huang CY, Lee JK, Chen ZW, Cheng JF, Chen SY, Lin LY, Wu CK. Inhaled Prostacyclin on Exercise Echocardiographic Cardiac Function in Preserved Ejection Fraction Heart Failure. Med Sci Sports Exerc. 2020 Feb;52(2):269-277. doi: 10.1249/MSS.0000000000002145. PMID 31479003